CLINICAL TRIAL: NCT03506867
Title: A Healthy People Initiative (HPI) - Community-Based Participatory Action Pragmatic Parallel Arm Multi-Site Randomized Controlled Trial Using The Bridge ModelTM in Systemically Disadvantaged Populations: HPI Trial Protocol
Brief Title: Healthy People Initiative (HPI)
Acronym: HPI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20180274-01H
Record Dates: First submitted 2018-03-29; First posted 2018-04-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Nicotine Dependence; Substance Use Disorders
Keywords: Health Equity; Community Based Participatory Action Research; Poverty Reduction
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The HPI study is a crossover, community-based, multi-site pragmatic RCT (1:1 allocation ratio) in Ottawa and Toronto. It uses a 12-month follow-up to evaluate short- and long-term effects of the intervention on health, social, and economic outcomes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research staff analyzing the data will be blinded to the allotment and reported outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care arm (Active Comparator): We will provide the participants in this arm with pamphlets and knowledge about available services in the city through partner agencies.
  Interventions: Behavioral: Life skills, training, education and work/volunteer opportunities
- Life skills, training, education and work/volunteer opportunities, and peer support (Active Comparator): The life skills, training, education, work/volunteer opportunities, and peer support arm will be offered to the usual care arm participants after the first six months of study enrollment.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Life skills, training, education and work/volunteer opportunities — Intervention arm will receive proactive and sustained access to enhanced education and socio-economic supports (e.g. volunteer and/or work opportunities).
  Arms: Usual care arm
Behavioral: Usual Care — We will provide the participants in this arm with pamphlets and knowledge about available services in the city through partner agencies.
  Arms: Life skills, training, education and work/volunteer opportunities, and peer support

SUMMARY:
Addictions do not occur in isolation. Tackling addictions requires addressing social determinants such as isolation, homelessness, marginalization, and unemployment. Research on individuals living with or at risk for HIV/AIDS highlights that unemployment correlates with higher levels of depression, anxiety, and social isolation compared to employment. In Ottawa, the PROMPT project engaged homeless or at-risk populations, including people who use drugs and those living with or at risk for HIV/AIDS or Hepatitis C using the Bridge ModelTM, a pragmatic community-based participatory action research approach operationalized through earlier projects at the Bridge Engagement Center in Ottawa, Canada. The PROMPT project demonstrated that implementing multi-component, complex interventions is both feasible and effective, achieving broader socio-economic outcomes beyond reduction and quitting tobacco and poly-substance use. However, PROMPT participants identified a lack of social and recovery capital -family and social connections, opportunities for volunteering and jobs- as a major barrier to recovery. To address this, we conducted a six-month feasibility pilot study with 20 PROMPT participants. By its conclusion, 15 participants were engaged in small paid or volunteer roles, including educational opportunities, fostering both social integration and recovery. Insights from this pilot study informed the design of a larger community-based multi-site pragmatic randomized trial (RCT) to further evaluate the effectiveness of the Bridge ModelTM, the Healthy People Initiative (HPI) project. The Healthy People Initiative (HPI) is a community-based, participatory, pragmatic parallel-arm multi-site with a cross-over design, recruiting 250 participants (16+) at risk of homelessness or low socioeconomic status in Ottawa and Toronto, Canada.

DETAILED DESCRIPTION:
Title of Trial: A Healthy People Initiative (HPI) - Community-Based Participatory Action Pragmatic Parallel Arm Multi-Site Randomized Controlled Trial using The Bridge ModelTM in Systemically Disadvantaged Populations: HPI Trial Protocol

Short Title of Trial: HPI Trial

Principal Investigator: Smita Pakhalé

Trial Sites: Ottawa (The Bridge Engagement Centre) & Toronto (Parkdale Activity Recreation Centre)

Primary outcome: The Healthy People Initiative (HPI) randomized controlled trial (RCT) builds on the pilot study to evaluate changes in participants' self-reported quality of life (QoL) as the primary outcome while implementing the Bridge Model™ approach to address tobacco management.

Secondary outcomes: The secondary objective is to quantify reductions in tobacco use and quitting tobacco use altogether, with quit rates validated biochemically, and changes in self-efficacy.

Tertiary outcomes: These include evaluating process-related metrics such as participant enrolment rates, consent rates, and adherence to protocol; estimating implementation costs to guide future cost-effectiveness analyses; and assessing additional patient-reported outcomes such as self-efficacy, participation in education or employment, and reductions in polysubstance use. Additionally, a cost-utility analysis from a health system perspective will assess the economic impact of the 52-week intervention by measuring total costs and healthcare utilization, linking trial data to administrative health records. We aim to provide robust evidence to support the utility of the Bridge ModelTM in addressing health and social inequities through community-driven, peer-led interventions that integrate social determinants with individual health outcomes.

Primary Objective: To assess the feasibility of a randomized controlled trial investigating access to improvements in 'social capital' in the low income population in Ottawa and Toronto.

Study Design & Population: The HPI study is a crossover, community-based, multi-site pragmatic RCT (1:1 allocation ratio) in Ottawa and Toronto. It uses a 12-month follow-up to evaluate short- and long-term effects of the intervention on health, social, and economic outcomes. Data sources include self-reports, biochemical validation, and administrative health records

Sample Size: 250

Trial Arms: The HPI RCT has two arms: usual care and intervention (Figure 1). The intervention arm employs the Bridge ModelTM, offering life-skills workshops, social integration, peer guidance, system navigation (e.g., housing), and APN (Advanced Practice Nurse) or NP (Nurse Practitioner) counselling, including primary care, preventive services, and referrals. Both arms receive monthly follow-ups from peers and APN/NP. Usual care includes resource information and counselling, with an option to switch to the intervention arm after six months. All participants receive nicotine replacement therapy (NRT) for 12 months as needed.

Trial Duration: 12 months Follow-up Duration: 12 months

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 16 years or older, reside in Ottawa or Toronto,
* Have smoked tobacco in the past 7 days
* Identify as low socioeconomic status and/or at risk of homelessness, and be available for in-person follow-up for one year.

Exclusion criteria:

* Declining consent
* Any person who is in or planning on accessing addictions treatment (in-patient drug rehabilitation) in Ottawa or Toronto and hence will be unavailable for follow up
* Currently or recently (in the past 30 days) enrolled in any other smoking cessation program

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Quality of Life | 12 Months
  To assess the trend in self-reported quality of life using the European Quality of Life 5 Dimensions 5 Level Version.

SECONDARY OUTCOMES:
Self-Reported Efficacy | 12 months
  To estimate change in self-reported self-efficacy.
Tobacco use | 12 months
  To estimate self-reported reduced or quit tobacco use rate (corroborated with the measurement of exhaled Carbon Monoxide) and poly-substance use rate.

OTHER OUTCOMES:
Consent and Protocol Violation Rate | 12 months
  The consent rate of eligible participants and the rate of protocol violations resulting in cross contamination of the groups receiving study intervention
Healthcare Utilization Rate | 12 months
  To compare healthcare utilization (ER visits and hospitalizations) over one year before and after the study by linking the trial data to health administrative data available at the Institute for Clinical and Evaluative Sciences (ICES).
Access to Work, Training, and Volunteer Opportunities | 12 months
  To assess access to work, training, or volunteering positions using a self-reported online survey.
Costs of Poverty Reduction Intervention | 12 months
  To estimate the costs of poverty reduction intervention (life skills workshops, training, and education/volunteer/employment opportunities.
Average Recruitment Rate | 12 months
  To assess the ability of participating sites to enroll an average of 6 participants per month.
Poly-substance use rates | 12 months
  Reductions in polysubstance use (biochemically validated)

CONTACTS AND LOCATIONS:
Overall Officials: Smita Pakhalé, MD, MSc, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Bridge Engagement Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Upon request study de-identified data will be made available to interested and qualified researchers.
Time Frame: Upon request study de-identified data will be made available to interested and qualified researchers. No time frame necessary.
Access Criteria: No access criteria. De-identified raw data will be available upon request.